CLINICAL TRIAL: NCT07228494
Title: Comparative Study of Simulation Technologies for Use in Neonatal Resuscitation Training for Rural Hospitals
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MaineHealth (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Misty Melendi, Principal Investigator, Chair of Neonatology, MaineHealth
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2240996
Record Dates: First submitted 2025-11-04; First posted 2025-11-14 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-11

CONDITIONS: Interprofessional Education; Neonatal Resuscitation; Rural Health
Keywords: HoloBaby; Neonatal resuscitation; interprofessional education; medical education; neonatal readiness; technology development; mixed reality

STUDY DESIGN:
Intervention Model Description: randomized cluster non-inferiority clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HoloBaby Arm (Experimental): Participants in this arm will complete their simulations with the HoloBaby simulator technology
  Interventions: Other: HoloBaby Technology
- High-fidelity Arm (Active Comparator): Participants in this arm will complete their simulations with the traditional high-technology high-fidelity neonatal simulator
  Interventions: Other: High Fidelity Simulator Technology

INTERVENTIONS:
Other: HoloBaby Technology — The intervention will be utilizing HoloBaby technology for Neonatal Resuscitation Simulation Education.
  Arms: HoloBaby Arm
Other: High Fidelity Simulator Technology — The intervention will be utilizing HiFi simulator technology for Neonatal Resuscitation Simulation Education.
  Arms: High-fidelity Arm

SUMMARY:
Conduct a randomized cluster non-inferiority clinical trial with teams of interprofessional neonatal clinicians from rural delivery hospitals. In this trial we will compare HoloBaby, a novel mixed reality simulator technology, to traditional high-technology simulator technology.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age
* primary clinical role is either physicians, nurses, or respiratory therapists
* have completed NRP® certification within the two years prior to enrollment
* attend deliveries at participating hospital in study

Exclusion Criteria:

- chronic neck pain, a previous neck injury that requires ongoing precautions, severe motion sickness or vertigo, and/or photosensitive epilepsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2026-01-08 (Estimated); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Team-based NRP® Adherence Score | 13 months
  the change in resuscitation performance at each site over time; NRP score will be measured utilizing an NRP adherence assessment tool that has been published with validity evidence. the adherence score will be presented as a percentage (out of 100) and higher scores indicate a higher adherence to NRP guidelines thus indicating a better resuscitation performance

CONTACTS AND LOCATIONS:
Locations (1):
- MaineHealth Maine Medical Center Portland, Portland, Maine, United States

IPD SHARING:
Plan to Share IPD: No
data collected is team-based data